CLINICAL TRIAL: NCT04380584
Title: Relation Between Plasma Apelin Level and Diabetic Nephropathy in Type 2 Diabetic Patients
Brief Title: Relation Between Plasma Apelin Level and Diabetic Nephropathy in Type 2 Diabetes Patients.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Youssry Helmy, Lecturer of internal medicine, Cairo University
Other Study IDs: N-4-2020
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Diabetic Nephropathies
Keywords: Apelin; Type 2; Diabetes; Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples Without DNA — serum Apelin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- I: 30 patients with type 2 DM with nephropathy
  Interventions: Diagnostic Test: plasma Apelin level
- II: 30 type 2 DM without nephropathy
  Interventions: Diagnostic Test: plasma Apelin level
- III: 30 non DM as control group
  Interventions: Diagnostic Test: plasma Apelin level

INTERVENTIONS:
Diagnostic Test: plasma Apelin level — blood sample for detection of plasma Apelin level

SUMMARY:
Diabetic nephropathy (DN) is the commonest cause of chronic kidney disease, and proteinuria isn't determent factor for the end stage renal disease in diabetics. Apelin is adipokine and have a beneficial role in early prediction of diabetic nephropathy. Few studies were done about apelin in diabetes. Purpose of the study: to investigate the association between the apelinergic system and diabetic nephropathy.

DETAILED DESCRIPTION:
Introduction Type 2 Diabetes Mellitus is a metabolic syndrome associated with hyperglycemia due to defect in secretion or action of insulin or both. Long term hyperglycemia leads to complications of microvasculature involving the eyes, kidneys and nerves.

Diabetic nephropathy (DN) is the commonest cause of end-stage renal disease that may need hemodialysis up to renal transplantation with increased incidence of mortality. Without management, patients with diabetes worsen from micro albuminuria to frank proteinuria with more impairment of kidney functions. This worsening develops in both type 1 and type 2 diabetes.Previous studies have revealed major roles of different inflammatory molecules in the development of diabetic nephropathy, including acute phase reactants, inflammatory cytokines, adhesion molecules, and chemokines.

Previous studies have revealed major roles of different inflammatory molecules in the development of diabetic nephropathy, including acute phase reactants, inflammatory cytokines, adhesion molecules.

Apelin (APLN) is the endogenous ligand peptide which is encoded in humans by the APLN gene. It is presented widely in different organs as the heart, kidney, liver, fatty tissue, endothelium, plasma, gastrointestinal tract, brain and adrenals .Apelin has a major role in the pathophysiology of hypertension, heart failure, cardio-vascular disease, DM, and obesity. Apelin is found to be higher in type 2 diabetic patients than healthy subjects. It inhibits insulin secretion, so it may precipitates impaired metabolism of glucose.

Also, Apelin present in omental fat is higher than its presence in subcutaneous fat suggesting its contribution to central obesity which is an important risk factor for type 2 DM.

In diabetic nephropathy, the apelin-13 level is markedly higher in than non-diabetic organs. Apelin mediates podocyte apoptosis,that is inversely related with podocyte autophagy in nephropathic diabetic mice. In addition, the mTOR pathway is supposed to have responsibility for inhibiting podocyte autophagy by apelin.

Apelin participates in the pathology of glomerular angiogenesis by affecting the permeability in glomeruli and glomerular endothelial cells proliferation of diabetics. So, playing a role in DN pathogenesis. Also, administration of apelin-13 diabetic rats restored the down regulation of the antioxidant catalase, revealing its renal protective effect via antioxidant pathways.

We aimed from this work to evaluate the relation between plasma Apelin level and diabetic nephropathy in Egyptian Type 2 diabetic patients.

Materials and methods After approval by the research ethical committee of Kasr El Ainy faculty of medicine, Cairo University on research protocols. A case control study including 90 patients aged 20 to 65 years, 30 healthy subjects as a control group and 60 patients with type 2 DM .Patients were collected from the endocrinology outpatient clinic, Kasr El Ainy, Cairo university. It was conducted from November 2019 to march 2020.

Oral consent was obtained from patients before inclusion after explaining the study protocol. Patients were divided into 3 groups, (group I) 30 patients with type 2 DM with nephropathy, (group II) 30 type 2 DM without nephropathy and (group III) 30 non DM as control group. Exclusion criteria included Patients with nephropathy due to other causes than diabetes, hepatic, intrinsic renal or coronary artery disease, patients with diabetic neuropathy and retinopathy and hypertensive patient on angiotensin receptor blockers (ARBS) or angiotensin converting enzyme inhibitors (ACEI) treatment as it affect Apelin level.

Full medical history was taken from all subjects, emphasizing on age , duration of diabetes mellitus, complications specially nephropathy and other co-morbid conditions and full clinical examination including blood pressure measurement, weight, height, Body Mass Index (BMI) (kg/m2) and waist circumference .

Laboratory investigations in the form of fasting blood glucose (FBG), 2 hr- postprandial blood glucose (2 hr -PPG), fasting lipids {total cholesterol (TC), triglycerides (TAG), low densitylipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), glycosylated hemoglobin (Hb A1c), urea, creatinine, urine analysis , albumin creatinine ratio , estimated glomerular filtration rate (e GFR) , glycosylated hemoglobin (Hb A1c), and Apelin levels were assessed.

Sampling: Five ml of venous blood was collected by venipuncture was divided into 3 parts: The first part was 2 ml of blood added to a tube containing EDTA for determination of HbA1C by caution exchange resin. The 2nd part was 3 ml of blood was left in plastic serum tubes and the specimens were allowed to clot at room temperature then serum was separated from the cells as soon as by centrifugation at 3000xg for 5 minutes. The separated serum was stored at -20ºC until analysis. The 3rd part was collected in a tube containing EDTA and centrifuged for 15 min at 1000×g at 2-8℃ within 30 min of collection. The supernatant was collected and stored at -80ºC for apelin determination.

Determination of serum urea, serum creatinine, serum total cholesterol, serum triglyceride, serum LDL and serum HDL were carried out on Dimension RxL Max analyzer, (Siemens Healthcare GmbH - Henkestr. 127, 91052 Erlangen, Germany) by colorimetric techniques.

Plasma apelin was determined using competitive-ELISA kit supplied from Elabscience Biotechnology Inc., (1 Shizishan Street, Hongshan District, Wuhan, Hubei, China) , ( Estienne A et al . 2019). eGFR was estimated using Cockcroft Gault equation: Cockcroft Gault equation= 140-age x weight/72 x S.Cr mg/dl(x 0.85 in female).

Complete urine analysis was done to detect the presence of active urinary sediment (proteinuria, pyuria, RBCs or RBCs casts, granular cast).

Albumin concentrations were measured in urine using a Minineph micro albumin kit based on nephelometry method on Minineph-nephelometer. Urinary creatinine was determined on Dimension RxL Max analyzer by colorimetric technique and the ratio of urine albumin to creatinine was used to define micro albuminuria.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes patients of both sexes ,20-60 years of age

Exclusion Criteria:

* Patients with nephropathy due to other causes than diabetes, hepatic, intrinsic renal or coronary artery disease, patients with diabetic neuropathy and retinopathy and hypertensive patient on angiotensin receptor blockers (ARBS) or angiotensin converting enzyme inhibitors (ACEI)

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 90 patients aged 20 to 65 years, 30 healthy subjects as a control group and 60 patients with type 2 DM .Patients were collected from the endocrinology 84 outpatient clinic, Kasr El Ainy, Cairo university
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
prediction of diabetic nephropathy | 12 weeks
  the use of plasma apelin level as a predictor for development of diabetic nephropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
no sharing

REFERENCES:
- [Background] 1. American Diabetes Association (ADA) .2012. Diagnosis of diabetes mellitus.2012 .Diabetes 291 Care;35. suppl S64- S71. doi: 10.2337/dc12-s064 . 292 2. Bonnet F and Cooper ME. 2000. Potential influence of lipids in diabetic nephropathy:insights 293 from experimental data and clinical studies. Diabetes Metab.;26:254-64. 294 3. Chan YH. 2003: Biostatistics102: Quantitative Data - Parametric & Non-parametric Tests. 295 Singapore Med J.;44(8): 391-396. 296 4. Chan YH. 2003: Biostatistics 104: Correlational Analysis. Singapore Med J.;44(12) : 614- 297 619.